CLINICAL TRIAL: NCT01080898
Title: Evaluation of the Sensitivity and Specificity of Optical Coherence Tomography Combined With Fundus Color Photos for Diagnosis of Choroidal Neovessels in Age-related Macular Degeneration
Brief Title: Evaluation of Optical Coherence Tomography.
Acronym: ESSO
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: K080904; IDRCB 2009-A00670-57 (Other: AFSSAPS)
Record Dates: First submitted 2010-01-28; First posted 2010-03-04 (Estimated); Last update posted 2012-07-23 (Estimated); Status verified 2011-04

CONDITIONS: Age-Related Macular Degeneration; Choroidal Vessels; Anastomosis
Keywords: Age - Related Macular Degeneration; Optical Coherence Tomography; Choroidal neovascularization; FLORESCEIN Angiography; Fundus photographs
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- DMLA patients: patients > 50 years with suspicion of choroidal neo-vessels complicating age related macular degeneration (DMLA)
  Interventions: Other: tests

INTERVENTIONS:
Other: tests — color photographs, FLUORESCEIN angiography and OCT

SUMMARY:
Determination of the sensitivity and specificity of different combinations of imaging techniques (spectral domain optical coherence tomography, fundus photography and fluorescein angiography) used for the diagnosis of choroidal neovessels complicating age -related macular degeneration. This information will help to determine the choice of the most suitable combination for the above diagnosis.

DETAILED DESCRIPTION:
The following combinations will be studied: spectral domain optical coherence tomography (OCT) + fundus photography; fluorescein angiography + fundus photography and the combination of all three techniques (OCT+ fundus photography + fluorescein angiography).The sensitivity and specificity of the latter combination will be assessed by comparison with the results for this combination reported by several readers. Inter- and intra-observer reproducibility of the different combinations will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Age> 50 years
* First visit for suspicion of choroidal neo-vessels complicating age related macular degeneration
* Fundus color photographs , FLUORESCEIN angiography and OCT prescription

Exclusion Criteria:

* Age < 50 years
* Diabetes
* Central vein occlusion Macular hole Epi-retinal membrane Retinal detachment Macular hemorrhage more than the 1/3 of the lesion
* History of macular laser, PDT or intra-vitreal injection

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients > 50 years with suspicion of choroidal neo-vessels complicating age relatid macular degeneration (DMLA)
Sampling Method: Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2010-04; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of the sensitivity and specificity of optical coherence tomography combined with fundus color photos in the diagnosis of choroidal neovessels in age- related macular degeneration. | all outcome the day of inclusion

SECONDARY OUTCOMES:
Evaluation of the sensitivity and specificity of fluorescein angiography combined with fundus color photography in the diagnosis of choroidal neovessels in age - related macular degeneration. | all the outcome the day of inclusion
Evaluation of the sensitivity and specificity of optical coherence tomography combined with fundus color photography, and of fluorescein angiography combined with fundus color photography. | all outcome the day of inclusion
Rate of unusable images for each technique | all outcome the day of inclusion
Evaluation of the sensitivity and specificity of optical coherence tomography combined with fundus color photography for the diagnosis of sub-categories of choroidal neovessels | all outcome the day of inclusion
Evaluation of the sensitivity and specificity of fluorescein angiography combined with fundus color photography for the diagnosis of sub-categories of choroidal neovessels. | all outcome the day of inclusion
Evaluation of the intra-and inter-reader reproducibility of the diagnosis of choroidal neovessels in age-related macular degeneration using fluorescein angiography combined with fundus color photography. | all outcome the day of inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Ramin TADAYONI, MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris